CLINICAL TRIAL: NCT03660254
Title: Effect of Tai Chi on Functional Fitness of Elderly Patients With Degenerative Arthritis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chen Li Tien (Other)
Responsible Party: Sponsor-Investigator, Chen Li Tien, Research assistant, Taipei Medical University
Organization: Taipei Medical University (Other)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Health Services Research
Other Study IDs: b409103042@tmu.edu.tw
Record Dates: First submitted 2018-05-22; First posted 2018-09-06 (Actual); Last update posted 2018-09-06 (Actual); Status verified 2018-09

CONDITIONS: Exercise Training
MeSH Terms: interventions — Tai Ji

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- one group has exercise intervention (Experimental): tai chi exercise intervention，two times a week and each time costs one hour
  Interventions: Behavioral: tai chi
- no intervention (No Intervention): no intervention

INTERVENTIONS:
Behavioral: tai chi — tai chi exercise intervention，two times a week and each time cost one hour
  Arms: one group has exercise intervention

SUMMARY:
Degenerative arthritis is a common disease in the elderly , in recent years, there are young trends, the symptoms often cause great pain in the elderly, associated with lower physical exercise caused by decreased muscle mass, functional fitness performance Is also poor, affecting the ability of elderly people to live independently. Therefore, this study mainly explores whether the intervention of tai chi can improve the functional fitness of the elderly and reduce the pain index of the elderly. The study was designed to take the sample, which was divided into experimental group and control group. It was expected to receive 100 people. The subjects were asked to use the basic information, Karnofsky scale, The functional fitness test, the exercise conscious scale and the WOMAC pain scale were used as the research tools. The SPSS system was used to analyze whether the functional fitness index and the pain index were significantly different before and after exercise intervention. Whether the exercise intervention has an effect on the elderly.

DETAILED DESCRIPTION:
Degenerative arthritis is a common disease in the elderly , in recent years, there are young trends, the symptoms often cause great pain in the elderly, associated with lower physical exercise caused by decreased muscle mass, functional fitness performance Is also poor, affecting the ability of elderly people to live independently. Therefore, this study mainly explores whether the intervention of tai chi can improve the functional fitness of the elderly and reduce the pain index of the elderly. The study was designed to take the sample, which was divided into experimental group and control group. It was expected to receive 100 people. The subjects were asked to use the basic information, Karnofsky scale, The functional fitness test, the exercise conscious scale and the WOMAC pain scale were used as the research tools. The SPSS system was used to analyze whether the functional fitness index and the pain index were significantly different before and after exercise intervention. Whether the exercise intervention has an effect on the elderly.

ELIGIBILITY:
Inclusion Criteria:

1. Elderly persons aged 65 or above who actively participate in community activities
2. awareness MMSE score ≧ 25 and can use the Chinese, Taiwanese fluent communication
3. can stand for more than 60 minutes and the Kirsley scale for the second to zero level.

Exclusion Criteria:

1. medical advice for those who can not exercise
2. suffering from significant cardiovascular and heart disease
3. suffering from high blood pressure, asthma, diabetes
4. those suffering from skeletal muscle disease

Ages: 65 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 1 (Actual)
Dates: Start 2017-12-01 (Actual); Primary Completion 2018-02-28 (Actual); Study Completion 2018-02-28 (Actual)

PRIMARY OUTCOMES:
height | 1 min
  Measuring the height of the subject
Weight | 1 min
  Measuring the weight of the subject
Muscle strength | 1 min
  measuring how many times of "sit and down" can he do in 30 secs
Endurance | 2 mins
  measuring how many times can he do "knee pull-in" in 2 mins
Heart rate | 2 mins
  measuring heart rate before and after knee pull-in
Softness(sit and reach test) | 1 min
  sitting on the floor with legs stretched out straight ahead， With the palms facing downwards, and the hands on top of each other or side by side, the subject reaches forward along the measuring line as far as possible.
balance(One foot station) | 2 mins
  measuring how long can he stand in one foot
walking | 1 min
  walking for 10 meters and measuring how long participants take

CONTACTS AND LOCATIONS:
Locations (1):
- Laozhuang Popular activity center, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No